CLINICAL TRIAL: NCT04470271
Title: Effectiveness of Implementing a Strategy to Re-linkage to Care of Patients With Hepatitis C Who Were Lost to Follow-up
Brief Title: Re-linkage to Care of Patients With Hepatitis C
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Austral University, Argentina (Other)
Responsible Party: Principal Investigator, Maria Julia Cremona, Coordinator, Austral University, Argentina
Other Study IDs: CIE N° P 20-008
Record Dates: First submitted 2020-07-04; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Viral Hepatitis C
Keywords: viral infection; outcome; antiviral therapy
MeSH Terms: conditions — Hepatitis C; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients under routine hepatitis C care: Patients who are routinely followed at the treating institution. Investigators will evaluate baseline demographic, liver fibrosis stage, liver-related complications, and antiviral therapy.
- Patients with hepatitis C lost of follow-up: Patients who were lost of follow-up. Participants will be contacted to evaluate if the continued HCV care at another institution, were not routinely followed by a liver-specialist or if they died. Investigators will also evaluate baseline demographic, liver fibrosis stage, liver-related complications, and antiviral therapy.
  Interventions: Other: Patients with hepatitis C lost follow up

INTERVENTIONS:
Other: Patients with hepatitis C lost follow up — Patients with chronic HCV who were lost of follow up will be contacted by phone or email. At least 3 phone calls will be made on three different days. In case the patient is not contacted it will be considered lost of follow-up
  Groups: Patients with hepatitis C lost of follow-up

SUMMARY:
The purpose of this study is to identify patients with chronic hepatitis C virus (HCV) who were lost of follow up and relinkage them to hepatitis C care

DETAILED DESCRIPTION:
The investigators will review electronic medical charts to identify patients with HCV diagnosis. Next, investigators will evaluate if these patients are routinely followed by liver specialists at the Institution. Those patients who were lost of follow up will be reached to evaluate their disease and eventually offer them to restart HCV care.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients clinically evaluated at least once in the participating medical center
* chronic HCV infection

Exclusion Criteria:

* There are no exclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with history of chronic HCV infection who were lost of follow up.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who were lost of follow up | through study completion, an average of 6 months
  Participants are going to be contacted by phone or email to evaluate if they are under HCV care

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo O Silva, MD, Principal Investigator — Austral University, Argentina
Locations (1):
- Universidad Austral, Pilar, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No